CLINICAL TRIAL: NCT06932588
Title: Biomarker Role in Assessing Imaging Needs for Mild Cranial Trauma
Acronym: BRAIN-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Jonathan A. Grossberg, Professor of Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STUDY00008711; 2025P010295 (Other: Emory IRB)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Brain Injuries; Head Injury
Keywords: Biomarkers; Brain imaging; Brain trauma; Head CT scan; Mild traumatic brain injury (mTBI)
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Healthcare providers will be randomly assigned to either be blinded to the biomarker results or receive the results to guide their decision on ordering head CT imaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Published Biomarker Group (Experimental): Biomarker results are provided to the ED provider immediately and before the decision to order a head CT is made. A print-out of the results will be handed to the provider or uploaded to the epic platform.
  Interventions: Diagnostic Test: Biomarker Testing using the Alinity Whole-blood TBI biomarker i-STAT
- Blinded Biomarker Group (Active Comparator): Biomarker results are not disclosed during the decision-making process for cranial imaging.
  Interventions: Diagnostic Test: Biomarker Testing using the Alinity Whole-blood TBI biomarker i-STAT

INTERVENTIONS:
Diagnostic Test: Biomarker Testing using the Alinity Whole-blood TBI biomarker i-STAT — The i-STAT TBI cartridge is a point-of-care, whole-blood, biomarker-based assay that measures the level of biomarkers associated with brain injury in the bloodstream 24 hours after injury. Blood samples (5-10cc of whole blood) will be collected upon admission during a routine blood drawing in the ED. These samples will be tested using the iSTAT system for mild TBI biomarkers.
  In a subset of admitted patients, serial blood draws and iSTAT testing will be performed at 4, 8, 16, and 24 hours, depending on the patient's length of stay.
  Other Names: i-STAT TBI

SUMMARY:
This study aims to determine whether a blood test can help doctors decide when to use a head CT scan for patients with a mild head injury. Researchers are investigating whether the results from this blood test can aid in making better decisions about patient care and potentially reduce the need for imaging.

In this study, researchers will collect blood samples to assess whether this specific blood test can help doctors decide when head imaging is necessary following a head injury. The goal is to determine whether the use of this test can reduce the number of head imaging procedures performed in the emergency department (ED).

DETAILED DESCRIPTION:
The Biomarker Role in Assessing Imaging Needs for Mild Cranial Trauma (BRAIN-CT) study aims to determine whether immediate access to blood biomarker data can help doctors decide when a CT scan is necessary for patients with mild traumatic brain injury (mTBI). The study will also explore how biomarker data influences clinical outcomes, such as hospital stay duration, costs, and recovery. Additionally, it will identify specific patient groups where biomarker results may alter imaging decisions, assess the ability of biomarkers to predict worsening symptoms and develop predictive models to improve the accuracy of these tests compared to CT scans.

The study will enroll adults presenting with suspected mild traumatic brain injury (mTBI) in the emergency department at Grady Memorial Hospital. Minors, pregnant individuals, wards of the state, prisoners, and those with cognitive impairments will not be enrolled.

Participants will undergo blood-based biomarker testing upon ED presentation. Healthcare providers will be randomly assigned to either be blinded to the biomarker results or receive the results to guide their decision on ordering head CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Mild TBI, defined as Glasgow Coma Scale (GCS) score 13-15, presenting within 24 hours of injury
* No prior head imaging for the same incident
* Presenting within 24 hours of onset of injury

Exclusion Criteria:

* Patients with penetrating head injury
* History of known brain abnormality including tumor, cerebrovascular malformation, recent brain surgery (within 6 months), prior head injury (within 6 months)
* Need for emergent surgical intervention for brain or alternate body organ injury
* Need for emergent bedside procedures for hemodynamic or orthopedic stabilization
* Patients deemed at higher risk for decline by the provider prohibit the 15-minute delay in obtaining imaging needed for biomarker testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants having a CT head scan from biomarker positive | During hospital admission (average 15 days).
  The impact of biomarker results will be measured by the decision to obtain CT head imaging for patients presenting with mild TBI.

SECONDARY OUTCOMES:
Length of hospital stay | Hospital admission (average 15) days.
  Length of hospital stay until discharge
Number of participants with intracranial findings predicted by biomarker findings | Hospital admission (average 15) days.
  In participants undergoing CT head imaging, the proportion of participants with intracranial findings between biomarker-positive and biomarker-negative groups will be compared.
Number of readmissions for TBI-related symptoms | up to 6 months after hospital discharge
  Data will be taken from electronic medical records (EMR) and participant's interviews.
Glasgow Outcome Scale-Extended (GOS-E) | 6 months after hospital discharge
  Functional outcome measured by the GOS-E. The Glasgow Outcome Scale-Extended (GOS-E) is one of the most widely used outcome instruments to assess global disability and recovery after traumatic brain injury. The patient's overall rating is based on the lowest outcome category indicated on the scale. The overall rating is the lowest outcome category indicated by the person's answers (after discounting limitations or problems before injury). Deaths are taken from records, and on the GOS-E rating schema, a vegetative state (VS) or a score of 2 is the lowest category, and Upper Good Recovery (Upper GR) or a score of 8 is the highest. If the person has no limitations or impaired symptoms, their GOS-E rating is Upper GR (8).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grossberg, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share deidentified Individual participant data underlying the results reported in publications.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared starting 12 months and ending 3 years after the article's publication.
Access Criteria: Investigators with approved data use by an Institutional Review Board may submit proposals up to 3 years after the article's publication.

REFERENCES:
- [Derived] Tfaily A, Chacon A, Ma T, Ratcliff J, Smith R, Saad H, Reisner A, Gimbel D, Wang K, Kobeissy F, Grossberg JA, Alawieh AM. Biomarker role in assessing imaging needs for mild cranial trauma (BRAIN-CT): study protocol for a single-center, randomized controlled trial. Front Neurol. 2026 Jan 9;16:1692163. doi: 10.3389/fneur.2025.1692163. eCollection 2025. PMID 41586091